CLINICAL TRIAL: NCT04056065
Title: A Prospective, Multi-centric, Randomized, Double-blind, Parallel, Saline Controlled Phase II Safety and Efficacy Study of PMZ-2010 as a Resuscitative Agent for Hypovolemic Shock to be Used Along With Standard Shock Treatment.
Brief Title: PMZ-2010 (Centhaquine) as a Resuscitative Agent for Hypovolemic Shock
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Pharmazz, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PMZ-02 Version 03 2017; CTRI/2017/03/008184 (Registry Identifier: Clinical Trials Registry - India)
Record Dates: First submitted 2019-08-11; First posted 2019-08-14 (Actual); Last update posted 2019-08-14 (Actual); Status verified 2019-08

CONDITIONS: Hypovolemic Shock; Blood Loss
Keywords: Resuscitative agent; Vasopressor
MeSH Terms: conditions — Shock; Hemorrhage | interventions — Saline Solution; centhaquine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Normal Saline (Active Comparator): Hypovolemic shock patients will be provided the standard of care. Following randomization 100 ml (equal volume to experimental arm) of normal saline will be administered intravenously over 1 hour.
  Interventions: Drug: Normal Saline
- PMZ-2010 (centhaquine) (Experimental): Hypovolemic shock patients will be provided the standard of care. Following randomization PMZ-2010 (0.01 mg/kg) will be administered intravenously over 1 hour in 100 mL of normal saline.
  Interventions: Drug: Centhaquine

INTERVENTIONS:
Drug: Normal Saline — In addition to standard of care normal saline to be used as vehicle in the phase-II study to assess efficacy of PMZ-2010 as a resuscitative agent for hypovolemic shock
  Other Names: Vehicle
  Arms: Normal Saline
Drug: Centhaquine — In addition to standard of care PMZ-2010 to be used as an experimental drug in the phase-II study to assess its efficacy as a resuscitative agent for hypovolemic shock
  Other Names: PMZ-2010
  Arms: PMZ-2010 (centhaquine)

SUMMARY:
This is a prospective, multi-centric, randomized, double-blind, parallel, controlled phase-II efficacy clinical study of PMZ-2010 therapy in patients with hypovolemic shock.

Centhaquine is highly safe and well tolerated. Toxicological studies showed high safety margin in preclinical studies. Its safety and tolerability has been demonstrated in a human phase I study in 25 subjects (CTRI/2014/06/004647; NCT02408731).

DETAILED DESCRIPTION:
Centhaquine (previously used names, centhaquin and PMZ-2010; International Non-proprietary Name (INN) recently approved by WHO is centhaquine) has been found to be an effective resuscitative agent in rat, rabbit and swine models of hemorrhagic shock, it decreased blood lactate, increased mean arterial pressure, cardiac output, and decreased mortality. An increase in cardiac output during resuscitation is mainly attributed to an increase in stroke volume. Centhaquine acts on the venous α2B-adrenergic receptors and enhances venous return to the heart, in addition, it produces arterial dilatation by acting on central α2A-adrenergic receptors to reduce sympathetic activity and systemic vascular resistance.

Unlike presently used vasopressors, centhaquine increased mean arterial pressure by increasing stroke volume and cardiac output, and it decreased systemic vascular resistance. The most common adverse effects of vasopressors as a class include arrhythmias, fluid extravasation, and ischemia. Centhaquine does NOT act on beta-adrenergic receptors, and therefore the risk of arrhythmias is mitigated. It is NOT a vasopressor; however, it increases blood pressure and cardiac output by augmenting venous blood return to the heart and enhanced tissue perfusion by arterial dilatation. Enhancing tissue perfusion is a significant advantage over existing vasopressors.

ELIGIBILITY:
Inclusion Criteria:

* Adult males or females aged 18-70 years.
* Patients with Hypovolemic shock due to blood loss admitted to the emergency room or ICU with systolic blood pressure ≤ 90 mmHg at presentation and continue to receive standard shock treatment (endotracheal intubation; fluid resuscitation and vasopressors). Standard of care to be provided to the patients shall be the one used in the particular hospital setup.
* Body weight 45 kg - 85 kg.
* Female subject is either: (1) Not of childbearing potential, defined as postmenopausal for at least 1 year or surgically sterile (bilateral tubal ligation, bilateral oophorectomy or hysterectomy) or, (2) If of childbearing potential, agrees to use any of the following effective separate forms of contraception throughout the study, up to and including the follow-up visits: Condoms, sponge, foams, jellies, diaphragm or intrauterine device, or A vasectomised partner OR abstinence.

Exclusion Criteria:

* Terminal illness
* Development of any other terminal illness not associated with Hypovolemic shock due to blood loss during the 28 day observation period
* Patient with severe brain injury or with a Glasgow Coma Scale (GCS) < 8
* Type of injury is not known
* Inability to obtain intravenous access
* Known pregnancy
* Cardiopulmonary resuscitation (CPR) before randomization
* Presence of a do not resuscitate order
* Patient taking beta adrenergic antagonists
* Untreated tension pneumothorax
* Untreated cardiac tamponade
* Bilateral absent pupillary light reflex (both pupils fixed and dilated)
* Patient is participating in another interventional study
* Patients with systemic diseases which were already present before having trauma, such as: cancer, chronic renal failure, liver failure, decompensated heart failure or AIDS

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2017-05-29 (Actual); Primary Completion 2018-09-19 (Actual); Study Completion 2018-10-21 (Actual)

PRIMARY OUTCOMES:
Incidence of PMZ-2010 related adverse events | 28 days
  The primary objective of the study is to determine incidence of drug (PMZ-2010) related adverse events.

SECONDARY OUTCOMES:
Volume of fluid administered | 48 hours
  Total volume of fluid administered - Mean through 48 hours
Volume of blood products administered | 48 hours
  Total volume of blood products administered - Mean through 48 hours
Vasopressor(s) infused | 48 hours
  Amount of total vasopressor(s) infused - Mean through 48 hours
Doses of study drug | 48 hours
  Number of doses of study drug administered in first 48 hours post randomization
Change in systolic and diastolic blood pressure | 48 hours
  Change in systolic and diastolic blood pressure - Mean through 48 hours
Change in blood lactate level | 48 hours
  Change in blood lactate level - Mean through 48 hours
Change in base-deficit | 48 hours
  Change in Base-deficit - Mean through 48 hours
Change in platelet count | 48 hours
  Change in platelet count as part of coagulation parameters mean through 48 hours. Platelets are parts of the blood that helps the blood clot. Average platelet counts are 150,000 to 450,000 number of platelets per microliter.
Change in prothrombin time | 48 hours
  Change in prothrombin time as part of coagulation parameters mean through 48 hours. Prothrombin time (PT) is a blood test that measures the time it takes for the blood to clot. The average time range for blood to clot is about 10 to 14 seconds.
Change in international normalized ratio (INR) | 48 hours
  Change in international normalized ratio (INR) as part of coagulation parameters mean through 48 hours. The results of the prothrombin time test vary from laboratory to laboratory, therefore, a ratio called the international normalized ratio (INR) is calculated. It allows for differences in laboratories across the world so that test results become more relevant and can be compared. The average INR range is 0.8 to 1.1.
Change in fibrinogen | 48 hours
  Change in fibrinogen as part of coagulation parameters mean through 48 hours. Fibrinogen is a protein, specifically a clotting factor (factor I), that is essential for proper blood clot formation. The reference range for fibrinogen is 150-400 mg/dL
Change in Multiple Organ Dysfunction Syndrome Score | 28 days
  Change in Multiple Organ Dysfunction Syndrome Score (MODS) - Mean through 28 days. MODS is a 5 grade scale from 0 to 4, where 0 is the best and 4 is the worst outcome.
Change in Acute Respiratory Distress Syndrome | 28 days
  Change in Acute Respiratory Distress Syndrome (ARDS) - Mean through 28 days. ARDS will be determined using Murray Score for Acute Lung Injury which is based upon radiological findings, oxygenation status, ventilation status of the patient. A lower score of 0 is the best and about 2.5 is the worst outcome.
Change in Glasgow coma score | 28 days
  Change in Glasgow coma score (GCS) - Mean through 28 days. GCS is a 15 point scale to assess the level of consciousness of patients where less than 3 is comatose state and 15 is fully awake.
Stay in hospital, in ICU and/or on Ventilator | 28 days
  Days in hospital, in ICU and/or on Ventilator - Mean through 28 days
Incidence of mortality | 28 days
  Proportion of patients with all-cause mortality at 48 hours and 28 days

CONTACTS AND LOCATIONS:
Overall Officials: Anil Gulati, Study Chair — Pharmazz, Inc.
Locations (7):
- India (7):
  - Seven Star Hospital, Nagpur, Maha
  - KLE's Dr. Prabhakar Kore Hospital & Medical Research Centre, Belagavi
  - Post Graduate Institute of Medical Education and Research, Chandigarh
  - Institute of Postgraduate Medical Education & Research and SSKM Hospital, Kolkata
  - Dayanand Medical College & Hospital, Ludhiana
  - New Era Hospital & Research Institute, Nagpur
  - ORIANA Hospital, Varanasi

IPD SHARING:
Plan to Share IPD: No
Plan to publish the findings after completion of the study

REFERENCES:
- [Background] Kontouli Z, Staikou C, Iacovidou N, Mamais I, Kouskouni E, Papalois A, Papapanagiotou P, Gulati A, Chalkias A, Xanthos T. Resuscitation with centhaquin and 6% hydroxyethyl starch 130/0.4 improves survival in a swine model of hemorrhagic shock: a randomized experimental study. Eur J Trauma Emerg Surg. 2019 Dec;45(6):1077-1085. doi: 10.1007/s00068-018-0980-1. Epub 2018 Jul 13. PMID 30006694
- [Background] Papalexopoulou K, Chalkias A, Pliatsika P, Papalois A, Papapanagiotou P, Papadopoulos G, Arnaoutoglou E, Petrou A, Gulati A, Xanthos T. Centhaquin Effects in a Swine Model of Ventricular Fibrillation: Centhaquin and Cardiac Arrest. Heart Lung Circ. 2017 Aug;26(8):856-863. doi: 10.1016/j.hlc.2016.11.008. Epub 2016 Dec 19. PMID 28385449
- [Background] Papapanagiotou P, Xanthos T, Gulati A, Chalkias A, Papalois A, Kontouli Z, Alegakis A, Iacovidou N. Centhaquin improves survival in a swine model of hemorrhagic shock. J Surg Res. 2016 Jan;200(1):227-35. doi: 10.1016/j.jss.2015.06.056. Epub 2015 Jun 29. PMID 26216751
- [Background] Gulati A, Zhang Z, Murphy A, Lavhale MS. Efficacy of centhaquin as a small volume resuscitative agent in severely hemorrhaged rats. Am J Emerg Med. 2013 Sep;31(9):1315-21. doi: 10.1016/j.ajem.2013.05.032. Epub 2013 Jul 19. PMID 23871440
- [Background] Lavhale MS, Havalad S, Gulati A. Resuscitative effect of centhaquin after hemorrhagic shock in rats. J Surg Res. 2013 Jan;179(1):115-24. doi: 10.1016/j.jss.2012.08.042. Epub 2012 Sep 2. PMID 22964270
- [Background] Gulati A, Lavhale MS, Garcia DJ, Havalad S. Centhaquin improves resuscitative effect of hypertonic saline in hemorrhaged rats. J Surg Res. 2012 Nov;178(1):415-23. doi: 10.1016/j.jss.2012.02.005. Epub 2012 Apr 2. PMID 22487389
- [Result] Anil Gulati, Dinesh Jain, Nilesh Agrawal, Prashant Rahate, Soumen Das, Rajat Chowdhuri, Deba Dhibar, Madhav Prabhu, Sameer Haveri, Rohit Agarwal, Manish Lavhale. Clinical Phase II Results Of PMZ-2010 (centhaquin) As A Resuscitative Agent For Hypovolemic Shock. Critical Care Medicine Volume 47, Issue 1, Page 12.
- [Derived] Gulati A, Jain D, Agrawal NR, Rahate P, Choudhuri R, Das S, Dhibar DP, Prabhu M, Haveri S, Agarwal R, Lavhale MS. Resuscitative Effect of Centhaquine (Lyfaquin(R)) in Hypovolemic Shock Patients: A Randomized, Multicentric, Controlled Trial. Adv Ther. 2021 Jun;38(6):3223-3265. doi: 10.1007/s12325-021-01760-4. Epub 2021 May 10. PMID 33970455